CLINICAL TRIAL: NCT01979731
Title: Effects Job Rotation in the Prevention of Work Related Musculoskeletal Disorders: Cluster Randomized Trial
Brief Title: Effects Job Rotation in the Prevention of Work Related Musculoskeletal Disorders
Acronym: Jobrotation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Collaborators: Maria Luiza Caires Comper (Unknown)
Responsible Party: Principal Investigator, Rosimeire Simprini Padula, PhD. Clinical Professor, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 18170313500000064
Record Dates: First submitted 2013-10-17; First posted 2013-11-08 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Musculoskeletal Diseases
Keywords: Occupational health; Ergonomics; Environments; Prevention and Control
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Job rotation (Experimental): The intervention group will perform rotation function, switching between tasks with low, moderate and high ergonomic risk and different requests for ergonomic body region added to ergonomic guidelines.
  Interventions: Other: Guidelines ergonomics
- Guidelines Ergonomics (Active Comparator): Manual material handling Orientation posture Orientation furniture Orientation in general
  Interventions: Other: Job rotation

INTERVENTIONS:
Other: Job rotation — The intervention group will perform rotation function, switching between tasks with low, moderate and high ergonomic risk and different requests for ergonomic body region added to ergonomic guidelines.
  Arms: Guidelines Ergonomics
Other: Guidelines ergonomics — Orientation about manual material handling, posture, furniture, rest break and others in general.
  Arms: Job rotation

SUMMARY:
The objective this study is evaluated if job rotation (change works that function every to work hours)contributes to reduce absence from work to complaints musculoskeletal disorders. And:

* Improve general health status
* Improve musculoskelettal symptoms
* Improve work performance
* Decrease costs with absence

DETAILED DESCRIPTION:
This study is single-blinded RCT, whose aim is to evaluate the effect of the rotation function in the prevention of musculoskeletal disorders in industrial workers Methods: Participants will be recruited from employees a textile industry. The inclusion criteria are: employees age between 18 and 65 years and be able to read and understand the questionnaires. The number of working hours lost due to leave for sick leave due to illness of the musculoskeletal system and connective tissue (M Group International Classification of Diseases, ICD-10) is used to estimate the sample size. The average time lost during the last three months, in companies where the study was conducted is approximately 1,100 hours. Assume that interventions will enable a reduction of this number by 10%, ie, the groups will have a difference of 100 lost working hours, with a standard deviation of 250 hours. Will be considered a statistical power of 80%, α=0.05 and a follow-up loss of up to 15%. Thus, 116 workers are required per group. The productive sectors included in the study will be pre- stratified from the level of exposure to ergonomic risk factors. The sectors with similar demands will be grouped and randomly divided between the intervention group and the control group. The intervention group will perform rotation function, switching between tasks with low, moderate and high ergonomic risk and different requests for ergonomic body region added to ergonomic guidelines. The control group will receive only the ergonomic guidelines. Primary outcomes: Absence from work due to sick leave due to disease of the musculoskeletal system and connective tissue. Secondary outcomes are: musculoskeletal symptoms (Nordic Questionnaire and EVA), ergonomic risk factors (Quick exposure Check and Job Factors Questionnaire), psychosocial factors and fatigue (Need for Recovery Scale (NFR), general health status (WHOQOL-bref), physical activity level (Baecke Questionnaire), productivity with Work Performance Questionnaire (HPQ) and costs (incremental cost effectiveness ratio). Outcomes will be assessed at baseline and after 3 , 6 and 12 months . The information on the amount of hours lost by removal for medical leave will be recorded daily. Expected results: It is expected that interventions to reduce the occurrence of musculoskeletal disorders and consequent worker absenteeism due to sick leave, 100 hours of work lost. It is expected that the results obtained in this study may contribute to setting standards in the field of Occupational Health, as well as for decision making of professionals working in this area.

ELIGIBILITY:
Inclusion Criteria:

* Sectors workers with production lines that allow switching between different tasks and requests biomechanical exposure levels ergonomic risk. And work is carried out in production cells.

Exclusion Criteria:

* Sector workers whose production lines are automated or semi-automated, possessing the pace of work determined by machinery and that the work stoppage is not possible.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Decrease musculoskeletal absence from work. | After 6 months
  Absence from work due to sick leave due to disease of the musculoskeletal system and connective tissue

SECONDARY OUTCOMES:
Decrease Musculoskeletal symptoms | After 6 months
  Musculoskeletal symptoms (Nordic Questionnaire1 and EVA)

OTHER OUTCOMES:
Change Geral Health Condictions | After 6 months
  Psychosocial factors and fatigue (Need for Recovery Scale (NFR), general health status (WHOQOL-bref), physical activity level (Baecke Questionnaire)
Reduced Cost effectiveness | After 6 months
  Productivity (Work Performance Questionnaire (HPQ) and costs (incremental cost effectiveness ratio).

CONTACTS AND LOCATIONS:
Overall Officials: Rosimeire S Padula, PhD, Study Director — Universidade Cidade de São Paulo
Locations (1):
- Rosimeire Simprini Padula, Atibaia, São Paulo, Brazil

REFERENCES:
- [Background] Comper ML, Padula RS. The effectiveness of job rotation to prevent work-related musculoskeletal disorders: protocol of a cluster randomized clinical trial. BMC Musculoskelet Disord. 2014 May 22;15:170. doi: 10.1186/1471-2474-15-170. PMID 24885958
- [Derived] Comper MLC, Dennerlein JT, Evangelista GDS, Rodrigues da Silva P, Padula RS. Effectiveness of job rotation for preventing work-related musculoskeletal diseases: a cluster randomised controlled trial. Occup Environ Med. 2017 Aug;74(8):545-552. doi: 10.1136/oemed-2016-104077. Epub 2017 Mar 1. PMID 28250047
- See also: Paper Protocol — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4040481/